CLINICAL TRIAL: NCT04055181
Title: Influence of rTMS on Symptoms and Cognition in Patients With Psychiatric Disorders
Brief Title: Influence of rTMS on Symptoms and Cognitive Function in Patients With Psychiatric Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing HuiLongGuan Hospital (Other)
Responsible Party: Principal Investigator, Xiang Yang Zhang, Professor, Beijing HuiLongGuan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CASPsy2
Record Dates: First submitted 2019-07-14; First posted 2019-08-13 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Schizophrenia; Major Depressive Disorder
Keywords: schizophrenia; smoking; rTMS; major depressive disorder
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major; Smoking | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- rTMS in schizophrenia patients (Active Comparator): In active rTMS, 10 Hz stimulations over left DLPFC occurred at a power of 110% of motor threshold (MT) for 27-s intervals with 20s inter-train interval. 20 minutes were administered each day (Monday-Friday) for 4 consecutive weeks
  Interventions: Device: rTMS in schizophrenia patients
- rTMS in schizophrenia Controls (Sham Comparator): In sham rTMS, all procedures were identical to 10Hz Schizophrenia group except they were the non-magnetized steel cylinders, instead of cylindrical magnets, that were rotated.
  Interventions: Device: rTMS in schizophrenia Controls
- rTMS in major depressive disorders patients (Active Comparator): In active rTMS, 10 Hz stimulations over left DLPFC occurred at a power of 110% of MT for 27-s intervals with 20s inter-train interval. 20 minutes were administered each day (Monday-Friday) for 4 consecutive weeks
  Interventions: Device: rTMS in major depressive disorders patients
- rTMS in major depressive disorders controls (Sham Comparator): In sham rTMS, all procedures were identical to 10Hz depression group except they were the non-magnetized steel cylinders, instead of cylindrical magnets, that were rotated.
  Interventions: Device: rTMS in major depressive disorders controls

INTERVENTIONS:
Device: rTMS in schizophrenia Controls — all procedures were identical to "rTMS in schizophrenia patients" group except they were the non-magnetized steel cylinders, instead of cylindrical magnets, that were rotated.
  Arms: rTMS in schizophrenia Controls
Device: rTMS in schizophrenia patients — 10 Hz stimulations over left DLPFC occurred at a power of 110% of MT for 27-s intervals with 20s intertrain interval. 20 minutes were administered each day (Monday-Friday) for 4 consecutive weeks
  Arms: rTMS in schizophrenia patients
Device: rTMS in major depressive disorders controls — all procedures were identical to "rTMS in major depressive disorders patients" group except they were the non-magnetized steel cylinders, instead of cylindrical magnets, that were rotated.
  Arms: rTMS in major depressive disorders controls
Device: rTMS in major depressive disorders patients — 10 Hz stimulations over left DLPFC occurred at a power of 110% of MT for 27-s intervals with 20s intertrain interval. 20 minutes were administered each day (Monday-Friday) for 4 consecutive weeks
  Arms: rTMS in major depressive disorders patients

SUMMARY:
The investigators investigated the effects of high frequency (10Hz) repetitive transcranial magnetic stimulation (rTMS) on the symptoms and cognitive functioning in patients with psychiatric disorders

DETAILED DESCRIPTION:
OBJECTIVE: This study aimed to evaluate the efficacy of high-frequency rTMS over left dorsolateral prefrontal cortex in the treatment of symptoms and cognitive functioning in 200 chronic patients with schizophrenia and 200 patients with major depressive disorders

METHODS:

1. Clinical Trial：The study consists of 4 weeks of treatment.
2. Assess Procedures:

2.1 Primary Outcome Variable-Psychopathology: The psychopathology of patients was assessed by three clinical trained staff, who were blind to treatment protocols, using the Positive and Negative Syndrome Scale (PANSS) or DSM-IV for depression, and repeatable battery for the assessment of neuropsychological status(RBANS).Patients are interviewed at screening, at at baseline, 4 weeks, 16 weeks.

2.2 Side effects: The side effect rating scale (UKU) was used to assess the side effect at baseline, 4 weeks, and 16 weeks.

2.3 Weight gain measurement: weight gain every week

ELIGIBILITY:
Inclusion Criteria:

For Schizophrenia Patients:

* Diagnosis of schizophrenia by two senior psychiatrists
* Between 18 and 60 years and Han Chinese
* Duration of symptoms at least 12 months
* With unresolved negative symptoms (Negative scale of PANSS ≥20 and positive scale of PANSS < 24)
* Smoking

For Major Depressive Disorder Patients:

* Diagnosis of Major depressive disorder by two senior psychiatrists
* Between 18 and 60 years and Han Chinese
* Duration of symptoms at least 12 months
* Smoking

Exclusion Criteria:

* Documented disease of physical diseases including, but not limited to seizure, epilepsy, aneurysm brain tumor, and stroke, dementia, parkinson's disease, Huntington's disease, multiple sclerosis
* Acute, unstable and/or significant and untreated medical illness (e.g., infection, unstable diabetes, uncontrolled hypertension)
* Severe headache for unknown reasons and cardiovascular diseases, intracranial metals, pacemakers, severe and those receiving electroconvulsive therapy in the past 3 months
* Past history of autoimmune and allergies, hypertension, lung disease, diabetes or cerebrovascular disease), past history of neurological illness (head trauma with loss of consciousness for more than 5 minutes) or family history of epilepsy increasing the risk of seizures
* Education level less than 5 years by subject report
* Receiving or planning to start the psychotherapy during the rTMS treatment or past received psychotherapy 6 months before the current study
* Subjects who suffered from alcohol or illegal drug abuse/dependence

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 800 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
symptoms assessed on PANSS | 4 weeks
  The Positive and Negative Syndrome Scale is often shorted as PANSS. It is a well-characterized and well-applied measurement instrument that measures positive and negative syndromes, their differential and general severity of illness. The items on the PANSS are defined with increasing levels from 1 to 7, the greater the value appears, the severe the level is: 1 = absent, 2 = minimal, 3 = mild, 4 = moderate, 5 = moderate-severe, 6 = severe, and 7 = extreme. The PANSS score is finalized by summation of ratings across different items, the potential range for positive and negative scales are from 7 to 49 whereas the General Psychopathology Scale is ranged between 16 to 112.
cognitive functioning assessed on RBANS | 4 weeks
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) is a test for identifying and characterizing abnormal cognitive decline in the elders and examining neuropsychological disorders for younger adults. The RBANS is comprised of five domains, which are Immediate Memory, Visuospatial /Constructional, Language, Attention and Delayed Memory. Each of the five index is based on two subtests except Delayed memory index consisting of four subtests. The score from each index is scaled by the age group with the scaled score mean to be 100 and standard deviation equals to 15, then the total RBANS scored is summed up of these indexes with the same normal mean and standard deviation. The lower the RBANS score the patient receives, the grave cognitive declination appears.
major depressive disorders assessed on Diagnostic and Statistical Manual of Mental Disorders (DSM-V) | 4 weeks
  The classification of major depressive disorder has been updated in the Fifth Edition of Diagnostic and Statistical Manual of Mental Disorder (DSM-V). It is defined by the lifetime absence of mania and hypomania, as well as one or more major depressive episodes. DSM description includes the diagnostic classification, the diagnostic criteria sets and the descriptive text. The diagnostic classification represents the official list of mental disorder with diagnostic codes that used by all U.S. health care professionals. The diagnostic criteria, specifically, the criteria for major depressive disorder consists: five or more out of nine related symptoms, symptoms cause significant distress or impairment, episode has not attribute to any substance or medical condition, the absent of psychotic disorder, the absent of any manic or hypomanic episode. Last but not the least, the descriptive text provides information like diagnostic features, diagnostic measures and functional consequences.

SECONDARY OUTCOMES:
Side effect assessed on UKU | 4 weeks
  The Udvalg for Kliniske Under-sogelser (UKU) side effect rating scale is a clinician-rated assessment uses to capture the side effects of psychotropic drug doses.
  It consists three parts: The first part, the single symptom rating scale. The scoring level may varied on the individual items but the general scale remains the same principle: 0= not or doubtfully present, 1 = present to a mild degree, 2 = present to a moderate degree, 3 = present to a severe degree. The greater level indicate, the severe the symptom becomes. The second part is a global assessment, where as 0 refers to no effect and 3 represents side effects that interfere moderately with the patient's performance. The last component is a statement of the results that the patient's side effects have for following up the medication. The decision are listed as from 0, "no action", to 3, "discontinuation of drug or changes to another preparation". The larger the number appears, the greater demand of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Y Zhang, MD,PhD, Principal Investigator — Institute of Psychology, Chinese Academy of Sciences
Locations (6):
- China (6):
  - Chaohu Hospital of Anhui medical unviersity, Chaohu, Anhui
  - Zhongshan Third People's Hospital, Zhongshan, Guangdong
  - Wuhan Mental Health Center, Wuhan, Hubei
  - Ganzhou Third Hospital, Ganzhou, Jiangxi
  - Ningxia Mental Health Center, Ning’an, Ningxia
  - Xi'an Mental Health Center, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: No
Data with be available on request

REFERENCES:
- [Background] Kozak K, Sharif-Razi M, Morozova M, Gaudette EV, Barr MS, Daskalakis ZJ, Blumberger DM, George TP. Effects of short-term, high-frequency repetitive transcranial magnetic stimulation to bilateral dorsolateral prefrontal cortex on smoking behavior and cognition in patients with schizophrenia and non-psychiatric controls. Schizophr Res. 2018 Jul;197:441-443. doi: 10.1016/j.schres.2018.02.015. Epub 2018 Feb 24. PMID 29486960
- [Background] Prikryl R, Ustohal L, Kucerova HP, Kasparek T, Jarkovsky J, Hublova V, Vrzalova M, Ceskova E. Repetitive transcranial magnetic stimulation reduces cigarette consumption in schizophrenia patients. Prog Neuropsychopharmacol Biol Psychiatry. 2014 Mar 3;49:30-5. doi: 10.1016/j.pnpbp.2013.10.019. Epub 2013 Nov 6. PMID 24211840
- [Background] Huang W, Shen F, Zhang J, Xing B. Effect of Repetitive Transcranial Magnetic Stimulation on Cigarette Smoking in Patients with Schizophrenia. Shanghai Arch Psychiatry. 2016 Dec 25;28(6):309-317. doi: 10.11919/j.issn.1002-0829.216044. PMID 28638206
- [Background] Zvolensky MJ, Bakhshaie J, Sheffer C, Perez A, Goodwin RD. Major depressive disorder and smoking relapse among adults in the United States: a 10-year, prospective investigation. Psychiatry Res. 2015 Mar 30;226(1):73-7. doi: 10.1016/j.psychres.2014.11.064. Epub 2014 Dec 9. PMID 25650047
- [Background] Benadhira R, Thomas F, Bouaziz N, Braha S, Andrianisaina PS, Isaac C, Moulier V, Januel D. A randomized, sham-controlled study of maintenance rTMS for treatment-resistant depression (TRD). Psychiatry Res. 2017 Dec;258:226-233. doi: 10.1016/j.psychres.2017.08.029. Epub 2017 Aug 18. PMID 28844559